CLINICAL TRIAL: NCT05547854
Title: Finalizing and Testing an Online Therapist Training and Assistance Program to Facilitate Implementation of Comprehensive Behavioral Intervention for Tic Disorders
Brief Title: Evaluation of an Online Comprehensive Behavioral Intervention for Tics (CBIT) Therapist Training Program
Acronym: CBIT-Trainer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Collaborators: Marquette University (Other); PsycTech, LLC (Unknown)
Responsible Party: Principal Investigator, Mike Himle, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00158298
Record Dates: First submitted 2022-09-02; First posted 2022-09-21 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Tics; Tic Disorders; Tourette Syndrome
Keywords: Comprehensive Behavioral Intervention for Tics
MeSH Terms: conditions — Tics; Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: Effectiveness-implementation hybrid non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be masked to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Therapist Training (Active Comparator)
  Interventions: Behavioral: Behavior Therapy Training Institute
- Online Therapist Training (Experimental)
  Interventions: Behavioral: CBIT-Trainer

INTERVENTIONS:
Behavioral: Behavior Therapy Training Institute — In-person therapist training will follow the Tourette Association of America's established Behavior Therapy Training Institute procedures and will consist of 12 hours of in-person training conducted over the course of 2 days. Day 1 will involve standardized didactic lectures on tic disorders and video demonstrations of therapeutic techniques. Day 2 will involve break-out groups and role-play practice of CBIT techniques. Participants (therapists) will receive up to three, 30-minute follow-up consultations with a training instructor while providing CBIT to a study-enrolled patient.
  Arms: In-Person Therapist Training
Behavioral: CBIT-Trainer — In the online therapist training condition participants will be provided with access to the CBIT-Trainer program and asked to complete the training over the course of 4 weeks. CBIT-Trainer is designed for the average user to complete in approximately 12 hours. Participants (therapists) will receive up to three, 30-minute follow-up consultations with a CBIT expert while providing CBIT to a study-enrolled patient.
  Arms: Online Therapist Training

SUMMARY:
Tic disorders are a class of childhood-onset neuropsychiatric disorders that occur in 1-3% of the population. Studies have shown that a non-drug treatment known as Comprehensive Behavioral Intervention for Tics (CBIT) is more effective than supportive therapy for reducing tics in children and adults. Although CBIT is now recommended as a first-line intervention for tic disorders, many patients do not have access to CBIT, in part due to a lack of trained therapists. Currently, the only option available for training therapists in CBIT is an intensive, two day, in-person behavior therapy training institute (BTTI). This study will compare the traditional in-person training approach to a recently developed online, self-paced CBIT therapist training program called CBIT-Trainer with regard to (1) therapists' ability to accurately administer CBIT and (2) change in the severity of patients' tic symptoms after being treated by a CBIT-trained therapist.

DETAILED DESCRIPTION:
Tic disorders are a class of childhood-onset neuropsychiatric disorders that occur in 1-3% of the population and often cause significant impairment in physical, social, academic, and interpersonal functioning and reduced quality of life. There is currently no cure for tic disorders, however large-scale randomized controlled trials have shown that a non-drug treatment known as Comprehensive Behavioral Intervention for Tics (CBIT) is more effective than supportive psychotherapy for reducing tics in both children and adults. Although CBIT is now recommended as a first-line intervention for tic disorders, many patients do not have access to CBIT, in part due to a lack of trained therapists. Given the need and desire for CBIT among individuals with tic disorders, high demand for therapist trainings, and the lack of therapists adequately trained in CBIT, there is a clear need for innovative ways to train more providers in this evidence-based treatment. To address this gap, the investigators recently developed an innovative online program for training therapists to deliver CBIT (called CBIT-Trainer). This study will test CBIT-Trainer against an intensive in-person therapist training program in a randomized controlled trial. This study will accomplish four aims: (1) to compare CBIT-Trainer to traditional in-person training on therapists' ability to administer CBIT with fidelity, (2) to compare CBIT-Trainer to in-person training on patient outcomes when patients are treated by a CBIT-trained therapist, (3) to identify therapist factors that might improve (or limit) adoption and use of CBIT-Trainer, and (4) to identify therapist factors likely to influence continued use of CBIT after training. These aims will be tested using an effectiveness-implementation hybrid randomized controlled trial comparing CBIT-Trainer (online therapist training) to the Tourette Association of America's Behavior Therapy Training Institute (in-person therapist training), which is the current gold-standard for training CBIT therapists. Therapist-patient dyads will be recruited to participate. The primary therapist outcome will be therapists' skill in delivering CBIT in a standardized role-play, which will be assessed at post-training (Week 0), after administering CBIT with a patient (Week 10), and at 6-month follow-up (Week 24). The primary patient outcome will be overall clinical improvement, which will be assessed at pre-treatment (Week 0), post-treatment (Week 10), and 6-month follow up (Week 24). Secondary therapist outcomes that will be assessed include changes in knowledge of tic disorders and CBIT; changes in comfort and self-efficacy in delivering CBIT; adherence to the CBIT protocol when treating a patient with tics; attitudes toward evidence-based practice and CBIT; and therapists' ratings of the acceptability, appropriateness, and feasibility of the training. Secondary patient outcomes that will be assessed include changes in motor and/or vocal tic severity; changes in overall psychological/behavioral, physical, and social functioning; and satisfaction with the treatment received.

ELIGIBILITY:
This study will recruit therapist-patient dyads who meet the criteria below:

Therapist Inclusion Criteria:

1. Have the equivalent of a Master's degree (or higher) in a mental/behavioral health, medical, or related discipline.
2. Professionally licensed or certified to practice in their area of speciality.
3. Attest that providing comprehensive behavioral intervention for tics (CBIT) to treat children and/or adults with tic disorders falls within their scope of practice according to state licensing laws and regulations in the therapist's jurisdiction.
4. Have never attended the Tourette Association of America's Behavior Therapy Training Institute or an equivalent focused on CBIT.
5. Have access to a secure personal computer with high-speed internet access.
6. Speaks fluent English.
7. Has identified, or is willing to try to identify, at least 1 child or adult patient with a tic disorder who meets the patient inclusion criteria and who might be willing to participate in the study as a member of the therapist-patient dyad, and for whom the therapist is licensed or certified to treat with CBIT according to state licensing laws and regulations in the therapist's jurisdiction.
8. Is willing to be randomly assigned to training condition.
9. Is willing, able, and has the necessary resources to travel to, and attend, one of several in-person training sites if assigned to the in-person training condition.

Therapist Exclusion Criteria:

(1) Therapist is a first, second, or third degree biological relative, stepparent, or legal guardian of the study-matched patient.

Patient Inclusion Criteria:

1. 7 years of age or older (with consenting adult for minors).
2. Self- or parent-reported diagnosis of a tic disorder (e.g., provisional tic disorder, persistent motor/vocal tic disorder, or Tourette's disorder) issued by a qualified professional.
3. Currently engages in at least one motor and/or vocal tic multiple times per day.
4. Patient (and consenting adult for minors) speaks fluent English.
5. Access to a private computer with high-speed internet access.

Patient Exclusion Criteria:

1. Patients will be excluded if the study team is unable to identify and enroll a patient-matched therapist who meets the therapist inclusion criteria.
2. Patient is a first, second, or third degree biological relative of the study-matched therapist or if the study-matched therapist is the patient's legal guardian.
3. Any serious psychiatric or neurological condition that requires more immediate intervention or would interfere with study participation, based on the assessment of the treating therapist or the study investigators.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Therapist scores on the CBIT Fidelity Checklist and Rating Scale at post-training | up to 2 weeks post-training
  The CBIT Fidelity Checklist and Rating Scale measures therapists' accuracy in administering 12 core components of CBIT during a standardized role-play. Items are rated using a series of 5-point Likert-type ratings ranging from "poor" to "excellent." Item ratings are aggregated to provide an overall fidelity rating ranging from 0-48. Higher ratings indicate better performance.
Therapist scores on the CBIT Fidelity Checklist and Rating Scale at post-treatment | 10-12 weeks post-training
  The CBIT Fidelity Checklist and Rating Scale measures therapists' accuracy in administering 12 core components of CBIT during a standardized role-play. Items are rated using a series of 5-point Likert-type ratings ranging from "poor" to "excellent." Item ratings are aggregated to provide an overall fidelity rating ranging from 0-48. Higher ratings indicate better performance.
Therapist scores on the CBIT Fidelity Checklist & Rating Scale at 6-month follow-up | 24-26 weeks post-training
  The CBIT Fidelity Checklist and Rating Scale measures therapists' accuracy in administering 12 core components of CBIT during a standardized role-play. Items are rated using a series of 5-point Likert-type ratings ranging from "poor" to "excellent." Item ratings are aggregated to provide an overall fidelity rating ranging from 0-48. Higher ratings indicate better performance.
Proportion of treatment responders at post-treatment on the Clinical Global Impression Improvement Scale (CGI-I) | 10-12 weeks from the start of treatment (post-treatment)
  The CGI-I is a single-item clinical rating of symptom improvement relative to baseline. Ratings on the CGI-I range from 1 (very much improved) to 7 (very much worse). CGI-I ratings of 1 (very much improved) or 2 (much improved) indicate positive treatment response. Higher scores are related to worse treatment response.
Proportion of treatment responders at follow-up on the Clinical Global Impression Improvement Scale (CGI-I) | 24-26 weeks from the start of treatment (6-month follow-up)
  The CGI-I is a single-item clinical rating of symptom improvement relative to baseline. Ratings on the CGI-I range from 1 (very much improved) to 7 (very much worse). CGI-I ratings of 1 (very much improved) or 2 (much improved) indicate positive treatment response. Higher scores are related to worse treatment response.
Patient changes in overall symptom severity on the Clinical Global Impression Severity Scale (CGI-S) | Up to 2 weeks prior to starting treatment (baseline), 10-12 weeks from the start of treatment (post-treatment), 24-26 weeks from the start of treatment (6-month follow-up)
  The CGI-S is a single-item clinical rating of the participant's illness at the time of the assessment. Ratings on the CGI-S range from 1 (slight psychiatric illness) to 7 (extremely severe psychiatric illness). Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Therapist change scores on the Tic Disorder & CBIT Knowledge Test | Up to 2 weeks pre-training and up to 2 weeks post training
  The Tic Disorder & CBIT Knowledge Test is a 20-item pre-post multiple choice test that assesses therapists' knowledge of several essential concepts taught during the psychoeducation component of CBIT. Scores are based on the percentage of items answered correctly. Higher scores indicate greater understanding and mastery of the material.
Therapist changes in self-efficacy to treat tic disorders as measured by the Therapist Self-Assessment & Rating Form | Up to 2 weeks pre-training, up to 2 weeks post-training, 10-12 weeks from the start of treatment delivery with a patient, 24-26 weeks from the start of treatment delivery with a patient
  The Therapist Self-Assessment & Rating Form is a therapist self-rating form developed for this study. It is a face-valid measure designed to assess therapists' self-efficacy regarding to their ability to competently and effectively treat tic disorders using CBIT and intent to use CBIT to treat tic disorders in the future. Ten self-statements are each rated on a 5-point Likert-type scale ranging from "Strongly Disagree" to "Strongly Agree." Higher scores indicate higher self-efficacy on each item.
Patient changes in tic severity as measured by the Yale Global Tic Severity Scale (YGTSS) Total Tic Score | Up to 2 weeks prior to starting treatment (baseline), 10-12 weeks from the start of treatment (post-treatment), 24-26 weeks from the start of treatment (6-month follow-up)
  The YGTSS is a clinician-rated interview assessing motor and vocal tics symptom severity during the past week. Motor and vocal tics are rated separately across 5 domains: number (0-5), frequency (0-5), intensity (0-5), complexity (0-5), and interference (0-5). The ratings for each motor and vocal tic domain are then summed to produce an overall total tic score ranging from 0-50 with higher scores indicating greater severity.
Patient changes in tic-related impairment as measured by the Yale Global Tic Severity Scale (YGTSS) Overall Tic Related Impairment Scores | Up to 2 weeks prior to starting treatment (baseline), 10-12 weeks from the start of treatment (post-treatment), 24-26 weeks from the start of treatment (6-month follow-up)
  The YGTSS Overall Tic Related Impairment Score is a single-item clinician rating of overall impairment caused by tics. Impairment is rated on a 0-50 scale with higher scores indicating greater impairment.
Patient treatment satisfaction scores on the Treatment Satisfaction Questionnaire (TSQ) at post-treatment | 10-12 weeks from the start of treatment (post-treatment)
  The TSQ is a brief 10-item self-report measure that assesses patients' satisfaction with their therapist and the treatment that they received. Each item is rated on a 4-point Likert-type scale. Scores range from 0-40 with higher scores indicating greater overall treatment satisfaction.
Patient treatment satisfaction on the Treatment Satisfaction Questionnaire (TSQ) at follow-up | 24-26 weeks from the start of treatment (6-month follow-up)
  The TSQ is a brief 10-item self-report measure that assesses patients' satisfaction with their therapist and the treatment that they received. Each item is rated on a 4-point Likert-type scale. Scores range from 0-40 with higher scores indicating greater overall treatment satisfaction.
Changes in psychological/behavioral symptoms and adaptive functioning as indicated by change scores on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric/Parent Proxy Profile 25 (for child patients & caregivers only) | Up to 2 weeks prior to starting treatment (baseline), 10-12 weeks from the start of treatment (post-treatment), 24-26 weeks from the start of treatment (6-month follow-up)
  The PROMIS Pediatric/Parent Proxy Profile 25 contains a collection of 25 caregiver and child-report items assessing psychological/behavioral symptoms in children in the following domains: anxiety, depressive symptoms, fatigue, pain interference, physical function-mobility, and peer relationships. Each item is rated on a 1-5 scale with higher scores indicate more severe symptoms or poorer adaptive functioning.
Changes in psychological/behavioral symptoms and adaptive functioning as indicated by change scores on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Profile (for adult patients only) | Up to 2 weeks prior to starting treatment (baseline), 10-12 weeks from the start of treatment (post-treatment), 24-26 weeks from the start of treatment (6-month follow-up)
  The PROMIS-29 Profile contains a collection of 29 patient-report items assessing psychological/behavioral symptoms in adults in the following domains: anxiety, depression, fatigue, pain interference, physical function, and ability to participate in social roles and activities. Each item is rated on a 1-5 scale with higher scores indicate more severe symptoms or poorer adaptive functioning. Higher scores indicate more severe symptoms or poorer adaptive functioning.

OTHER OUTCOMES:
Therapist change scores on the Evidence-Based Practice and Attitudes Scale (EBPAS) | Immediately pre- and post-training, 10-12 weeks from the start of treatment delivery with a patient, 24-26 weeks from the start of treatment delivery with a patient
  The EBPAS is a measure of providers' attitudes toward the adoption evidence-based interventions and has been shown to predict implementation outcomes such as initiation and sustained use of evidence-based interventions. It contains 15 items regarding the respondent's feelings about using new types of therapy, interventions, or treatments. Respondents rate the extent to which they agree with each item using a 5-point Likert-type scale ranging from "Not at all" to "To a Very Great Extent." Scores range from 0-75 with higher scores indicating more positive attitudes toward evidence-based practice.
Therapist scores on the Acceptability of Intervention Measure (AIM) at post-training | Immediately post-training
  The Acceptability of Intervention Measure (AIM) is a psychometrically validated measure of an intervention's acceptability. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater acceptability of the intervention.
Therapist scores on the Acceptability of Intervention Measure (AIM) at post-treatment | 10-12 weeks from the start of treatment delivery with a patient
  The Acceptability of Intervention Measure (AIM) is a psychometrically validated measure of an intervention's acceptability. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater acceptability of the intervention.
Therapist scores on the Acceptability of Intervention Measure (AIM) at follow-up | 24-26 weeks from the start of treatment delivery with a patient
  The Acceptability of Intervention Measure (AIM) is a psychometrically validated measure of an intervention's acceptability. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater acceptability of the intervention.
Therapist scores on the Intervention Appropriateness Measure (IAM) at post-training | Immediately post-training
  The Intervention Appropriateness Measure (IAM) is a psychometrically validated measure of an intervention's appropriateness for addressing a clinical problem or disorder. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater appropriateness of the intervention.
Therapist scores on the Intervention Appropriateness Measure (IAM) at post-treatment | 10-12 weeks from the start of treatment delivery with a patient
  The Intervention Appropriateness Measure (IAM) is a psychometrically validated measure of an intervention's appropriateness for addressing a clinical problem or disorder. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater appropriateness of the intervention.
Therapist scores on the Intervention Appropriateness Measure (IAM) at follow-up | 24-26 weeks from the start of treatment delivery with a patient
  The Intervention Appropriateness Measure (IAM) is a psychometrically validated measure of an intervention's appropriateness for addressing a clinical problem or disorder. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater appropriateness of the intervention.
Therapist scores on the Feasibility of Intervention Measure (FIM) at post-training | Immediately post-training
  The Feasibility of Intervention Measure (FIM) is a psychometrically validated measure of an intervention's feasibility for implementation. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater feasibility of the intervention.
Therapist scores on the Feasibility of Intervention Measure (FIM) at post-treatment | 10-12 weeks from the start of treatment delivery with a patient
  The Feasibility of Intervention Measure (FIM) is a psychometrically validated measure of an intervention's feasibility for implementation. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater feasibility of the intervention.
Therapist scores on the Feasibility of Intervention Measure (FIM) at follow-up | 24-26 weeks from the start of treatment delivery with a patient
  The Feasibility of Intervention Measure (FIM) is a psychometrically validated measure of an intervention's feasibility for implementation. It contains 4 items that are rated on a 1-5 scale ranging from "Completely Disagree" to "Completely Agree." Items are averaged to produce an overall score ranging from 1-5 with higher scores indicating greater feasibility of the intervention.
Number of patients reporting adverse events | Post-treatment (week 10) & 6-month follow-up (week 24)
  All health complaints, recent illness or injury, or need for medical consultation occurring since the baseline assessment will be recorded via a patient interview at post-treatment and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mouton-Odum, PhD, Principal Investigator — PsycTech, LLC; Michael Himle, PhD, Principal Investigator — University of Utah; Doug Woods, PhD, Principal Investigator — Marquette University
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Marquette University, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in any publication(s) may be provided to qualified researchers with academic interests in tic disorders and related conditions and expertise in the scoring and interpretation of the outcome measures administered. All data shared will be coded with no identifying information included. Approval of the request by the study primary investigators and execution of all applicable data sharing agreements are prerequisites to the sharing of data with the requesting party.

REFERENCES:
- [Background] Robertson MM. The prevalence and epidemiology of Gilles de la Tourette syndrome. Part 1: the epidemiological and prevalence studies. J Psychosom Res. 2008 Nov;65(5):461-72. doi: 10.1016/j.jpsychores.2008.03.006. Epub 2008 Oct 2. PMID 18940377
- [Background] Evans J, Seri S, Cavanna AE. The effects of Gilles de la Tourette syndrome and other chronic tic disorders on quality of life across the lifespan: a systematic review. Eur Child Adolesc Psychiatry. 2016 Sep;25(9):939-48. doi: 10.1007/s00787-016-0823-8. Epub 2016 Feb 15. PMID 26880181
- [Background] Conelea CA, Woods DW, Zinner SH, Budman CL, Murphy TK, Scahill LD, Compton SN, Walkup JT. The impact of Tourette Syndrome in adults: results from the Tourette Syndrome impact survey. Community Ment Health J. 2013 Feb;49(1):110-20. doi: 10.1007/s10597-011-9465-y. Epub 2011 Nov 4. PMID 22052430
- [Background] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Background] Wilhelm S, Peterson AL, Piacentini J, Woods DW, Deckersbach T, Sukhodolsky DG, Chang S, Liu H, Dziura J, Walkup JT, Scahill L. Randomized trial of behavior therapy for adults with Tourette syndrome. Arch Gen Psychiatry. 2012 Aug;69(8):795-803. doi: 10.1001/archgenpsychiatry.2011.1528. PMID 22868933
- [Background] Roessner V, Plessen KJ, Rothenberger A, Ludolph AG, Rizzo R, Skov L, Strand G, Stern JS, Termine C, Hoekstra PJ; ESSTS Guidelines Group. European clinical guidelines for Tourette syndrome and other tic disorders. Part II: pharmacological treatment. Eur Child Adolesc Psychiatry. 2011 Apr;20(4):173-96. doi: 10.1007/s00787-011-0163-7. PMID 21445724
- [Background] Pringsheim T, Doja A, Gorman D, McKinlay D, Day L, Billinghurst L, Carroll A, Dion Y, Luscombe S, Steeves T, Sandor P. Canadian guidelines for the evidence-based treatment of tic disorders: pharmacotherapy. Can J Psychiatry. 2012 Mar;57(3):133-43. doi: 10.1177/070674371205700302. PMID 22397999
- [Background] Pringsheim T, Holler-Managan Y, Okun MS, Jankovic J, Piacentini J, Cavanna AE, Martino D, Muller-Vahl K, Woods DW, Robinson M, Jarvie E, Roessner V, Oskoui M. Comprehensive systematic review summary: Treatment of tics in people with Tourette syndrome and chronic tic disorders. Neurology. 2019 May 7;92(19):907-915. doi: 10.1212/WNL.0000000000007467. PMID 31061209